CLINICAL TRIAL: NCT03796728
Title: LIPS: A Prospective, Open-label Study to Evaluate the Effectiveness of Juvéderm® VOLIFT™ With Lidocaine for Lip Augmentation
Brief Title: A Study to Evaluate the Effectiveness of Juvéderm® VOLIFT™ With Lidocaine for Lip Augmentation
Acronym: LIPS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CMO-MA-FAS-0512
Record Dates: First submitted 2018-12-17; First posted 2019-01-08 (Actual); Results first posted 2021-07-28 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Lip Augmentation

STUDY DESIGN:
Intervention Model Description: All participants will sign an informed consent form, and begin at the Screening Visit. Filler treatment (Juvéderm® VOLIFT™ with Lidocaine) will be performed at (Initial Treatment visit) and data will be collected at this visit for all relevant parameters as per the Schedule of Study Procedures, Treatments and Assessments. Fourteen days after the initial treatment, participants will return to the clinic and the Investigator will assess whether a Touch-up treatment is to be performed at this visit. Follow up visits will occur at Day 30 and 3, 6, and 12 months after the last treatment.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Juvéderm® VOLIFT™ with Lidocaine (Experimental): Initial treatment with Juvéderm® VOLIFT™ with Lidocaine injectable gel to augment the lips on Day 1, with an optional touch-up treatment 14 days later, if applicable. Volume was determined by the Investigator not to exceed 3.0 milliliters (mL).
  Interventions: Device: Juvéderm® VOLIFT™ with Lidocaine

INTERVENTIONS:
Device: Juvéderm® VOLIFT™ with Lidocaine — Injectable gel that is a sterile, biodegradable, non-pyrogenic, viscoelastic, clear, colorless, homogeneous gel implant (dermal filler).

SUMMARY:
This is an open-label, multi-center, study where eligible participants will undergo treatment with Juvéderm® VOLIFT™ with Lidocaine injected into the lips for lip augmentation.

DETAILED DESCRIPTION:
This is a prospective, open-label, multi-center, interventional, medical device, post-marketing study. Each participant will act as his/her own control. Eligible participants will undergo treatment with Juvéderm® VOLIFT™ with Lidocaine injected into the lips for lip augmentation.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18 years of age or older
* Signed the Institutional Independent Ethics Committee (IEC)-approved informed consent form prior to any study-related procedures being performed
* Accept the obligation not to receive any other facial procedures or treatments anywhere in the lower face (below the orbital rim), neck, and oral cavity at any time during the study that are not related to the study
* Women of childbearing potential must have a negative urine pregnancy test before each injectable treatment and practice a reliable method of contraception throughout the study
* Ability to follow study instructions and likely to complete all required visits and assessments, as assessed by the Investigator.

Exclusion Criteria:

* Has lip tattoos, piercings, facial hair, or scars that would interfere with visualization of the lips and perioral area
* Has dentures or any device covering all or part of the upper palate, and/or severe malocclusion or dentofacial or maxillofacial deformities
* Has undergone oral surgery (e.g., tooth extraction, orthodontia, or implantation) within 6 weeks before enrollment or is planning to undergo any of these procedures during the study
* Has ever undergone facial plastic surgery or received permanent facial implants (e.g., polymethylmethacrylate, silicone, polytetrafluoroethylene) anywhere in the face or neck, or is planning to be implanted with any of these products during the study
* Has undergone semi-permanent dermal filler treatment (e.g., hyaluronic acid, calcium hydroxylapatite, poly-L-lactic acid) in the lower face (below the orbital rim) within 24 months before enrollment or is planning to undergo such treatment during the study
* Has undergone mesotherapy or cosmetic resurfacing (laser, photo-modulation, intense pulsed light, radiofrequency, dermabrasion, chemical peel, or other ablative or non-ablative procedures) anywhere in the face or neck, or Botulinum toxin injections in the lower face (below the orbital rim) within 6 months before enrollment or is planning to undergo any of these procedures during the study
* Has used any lip plumping products within 10 days before enrollment or is planning to use such products during the study (study treatment may be delayed as necessary to accommodate this 10-day washout period)
* Has begun using any over-the-counter or prescription, oral or topical, anti-wrinkle products for the lips or around the mouth within 90 days before enrollment or is planning to begin using such products during the study (participants who have been on a regimen of such products for at least 90 days are eligible for the study if they intend to continue their regimen throughout the study)
* Is on an ongoing regimen of anti-coagulation therapy (e.g., warfarin) or non-steroidal anti-inflammatory drugs (NSAIDs) (e.g., aspirin, ibuprofen) or other substances known to increase coagulation time (e.g., herbal supplements with garlic or gingko) within 10 days of undergoing study device treatment (study treatment may be delayed as necessary to accommodate this 10-day washout period)
* Is on a concurrent regimen of lidocaine or structurally related local anesthetics (e.g., bupivacaine)
* Has a history of anaphylaxis, atopy, or allergy to lidocaine, hyaluronic acid (HA) products, or Streptococcal protein, or is planning to undergo desensitization therapy during the study
* Has an active inflammation, infection, cancerous or precancerous lesion, or unhealed wound in the mouth area
* Has porphyria
* Has epilepsy
* Has impaired cardiac conduction, severely impaired hepatic function, or severe renal dysfunction
* Has any uncontrolled disease
* Females who are pregnant, nursing, or planning a pregnancy
* Current enrollment in an investigational drug or device study, participation in such a study within 6 weeks before enrollment, or be planning to participate in another investigation during the course of this study
* Is an employee (or immediate relative of an employee) of the Investigator, Allergan, or a representative of Allergan

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-12-19 (Actual); Primary Completion 2020-06-09 (Actual); Study Completion 2020-06-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- Portugal (2):
  - Clinica Milenio, Lisbon
  - Clínica Secret Beauty, Lisbon
- United Kingdom (2):
  - Medical and Cosmetic Clinic, Edinburgh
  - MediZen Ltd, Sutton Coldfield

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Juvéderm® VOLIFT™ With Lidocaine
Started | 60
Completed | 36
Not Completed | 24
Not completed — Lost to Follow-up | 8
Not completed — Reason not Specified | 16

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set included all participants who were consented and enrolled into this study and were treated with the investigational product Juvéderm® VOLIFT™ with Lidocaine.
Arm/Group | Juvéderm® VOLIFT™ With Lidocaine
Number analyzed (Participants) | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.8 (9.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59
  Male | 1
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a ≥ 1-point Improvement (Increase) in the Lip Fullness Scale (LFS2) Compared to Baseline Assessment at Day 30
Description: The LFS2 is an Investigator assessment of overall lip fullness measured by a 5-point scale where: 0=Minimal (Flat or nearly flat contour; minimal red lip show), 1=Mild (Some red lip show; no lower lip pout), 2=Moderate (Moderate red lip show with slight lower lip pout), 3=Marked (Significant red lip show and lower lip pout), and 4=Very Marked (Very significant red lip show, lower lip pout, and upper lip pout). The percentage of participants with a ≥ 1-point Improvement (Increase) in the Lip Fullness Scale (LFS2) compared to Baseline are reported.
Time Frame: Baseline (Prior to Treatment) to Day 30
Population: Evaluable Set included all participants in the Full Analysis Set who had at least a Baseline and a Day 30 post-treatment efficacy assessment during the study.
Measure: Number; unit: percentage of participants
Arm/Group | Juvéderm® VOLIFT™ With Lidocaine
Number analyzed (Participants) | 59
percentage of participants | 93.2

2. Secondary Outcome: Number of Participants With Change From Baseline in the Investigator's Assessment of Oral Commissures Lines as Measured by the 4-point Oral Commissures Severity Scale (OCSS)
Description: The Investigator assessed the participant's oral commissures lines (lines at the corner of the mouth) using the OCSS 4 point scale where: 0=None (No wrinkle or fold; slight upturned corners), 1=Mild (Shallow, just perceptible wrinkle or crease; horizontal or slightly downturned corners), 2=Moderate (Moderately deep and/or long wrinkle or crease; downturned corners), and 3=Severe (Very deep and/or long wrinkle or crease; frown at rest). A negative change from Baseline indicates improvement. A positive change from Baseline indicates a worsening. The number of participants is reported for each of the following point changes from Baseline: -3 to 3 at each timepoint.
Time Frame: Baseline (Prior to Treatment) to Day 30, Months 3, 6, and 12
Population: Evaluable Set included all participants in the Full Analysis Set who had at least a Baseline and a Day 30 post-treatment efficacy assessment during the study. Number analyzed is the number of participants with available data for analysis at the given timepoint
Measure: Count of Participants; unit: Participants
Arm/Group | Juvéderm® VOLIFT™ With Lidocaine
Number analyzed (Participants) | 59
Participants
  Change from Baseline to Day 30: -3 Point Change | 0
  Change from Baseline to Day 30: -2 Point Change | 5
  Change from Baseline to Day 30: -1 Point Change | 29
  Change from Baseline to Day 30: 0 Point Change (No change) | 25
  Change from Baseline to Day 30: 1 Point Change | 0
  Change from Baseline to Day 30: 2 Point Change | 0
  Change from Baseline to Day 30: 3 Point Change | 0
  Change from Baseline to Month 3: number analyzed (Participants) | 52
  Change from Baseline to Month 3: -3 Point Change | 0
  Change from Baseline to Month 3: -2 Point Change | 4
  Change from Baseline to Month 3: -1 Point Change | 27
  Change from Baseline to Month 3: 0 Point Change (No change) | 21
  Change from Baseline to Month 3: 1 Point Change | 0
  Change from Baseline to Month 3: 2 Point Change | 0
  Change from Baseline to Month 3: 3 Point Change | 0
  Change from Baseline to Month 6: number analyzed (Participants) | 51
  Change from Baseline to Month 6: -3 Point Change | 1
  Change from Baseline to Month 6: -2 Point Change | 3
  Change from Baseline to Month 6: -1 Point Change | 22
  Change from Baseline to Month 6: 0 Point Change (No change) | 21
  Change from Baseline to Month 6: 1 Point Change | 4
  Change from Baseline to Month 6: 2 Point Change | 0
  Change from Baseline to Month 6: 3 Point Change | 0
  Change from Baseline to Month 12: number analyzed (Participants) | 36
  Change from Baseline to Month 12: -3 Point Change | 0
  Change from Baseline to Month 12: -2 Point Change | 3
  Change from Baseline to Month 12: -1 Point Change | 9
  Change from Baseline to Month 12: 0 Point Change (No change) | 22
  Change from Baseline to Month 12: 1 Point Change | 2
  Change from Baseline to Month 12: 2 Point Change | 0
  Change from Baseline to Month 12: 3 Point Change | 0

3. Secondary Outcome: Change From Baseline in Participant's Assessment of Overall Satisfaction With Lips as Measured by the FACE-Q Lips Questionnaire
Description: The FACE-Q™ is a validated 10 question assessment measuring how satisfied the participant is with their lips. Each question is answered on a 4-point scale where: 1=Very Dissatisfied, 2=Somewhat dissatisfied, 3=Somewhat satisfied, and 4= Very Satisfied. The responses to the items were converted to a 100-point Rausch transformed scale score: 0 (worst) to 100 (best). Higher scores indicate higher satisfaction. A positive change from Baseline indicates improvement.
Time Frame: Baseline (Prior to Treatment) to Day 30, Months 3, 6, and 12
Population: Evaluable Set included all participants in the Full Analysis Set who had at least a Baseline and a Day 30 post-treatment efficacy assessment during the study. Number analyzed is the number of participants with data available for analysis at the given timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Juvéderm® VOLIFT™ With Lidocaine
Number analyzed (Participants) | 59
score on a scale
  Change from Baseline to Day 30 | 45.2 (27.16)
  Change from Baseline to Month 3: number analyzed (Participants) | 52
  Change from Baseline to Month 3 | 42.7 (30.23)
  Change from Baseline to Month 6: number analyzed (Participants) | 51
  Change from Baseline to Month 6 | 38.5 (26.25)
  Change from Baseline to Month 12: number analyzed (Participants) | 36
  Change from Baseline to Month 12 | 23.6 (31.78)

4. Secondary Outcome: Number of Participants by Investigator's Assessment of Global Aesthetic Improvement Score Category as Measured by the 5-point Global Aesthetic Improvement Scale (GAIS)
Description: The Investigator assessed the participant's global aesthetic improvement using the GAIS 5-point scale where: 2=Much Improved, 1=Improved, 0=No Change, -1= Worse, and -2=Much Worse. The number of participants in each score response category at each timepoint is reported.
Time Frame: Day 30, Months 3, 6, and 12
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Juvéderm® VOLIFT™ With Lidocaine
Number analyzed (Participants) | 59
Participants
  Day 30: 2=Much Improved | 32
  Day 30: 1=Improved | 27
  Day 30: 0=No Change | 0
  Day 30: -1=Worse | 0
  Day 30: -2=Much Worse | 0
  Month 3: number analyzed (Participants) | 52
  Month 3: 2=Much Improved | 24
  Month 3: 1=Improved | 28
  Month 3: 0=No Change | 0
  Month 3: -1=Worse | 0
  Month 3: -2=Much Worse | 0
  Month 6: number analyzed (Participants) | 51
  Month 6: 2=Much Improved | 12
  Month 6: 1=Improved | 39
  Month 6: 0=No Change | 0
  Month 6: -1=Worse | 0
  Month 6: -2=Much Worse | 0
  Month 12: number analyzed (Participants) | 36
  Month 12: 2=Much Improved | 2
  Month 12: 1=Improved | 28
  Month 12: 0=No Change | 6
  Month 12: -1=Worse | 0
  Month 12: -2=Much Worse | 0

5. Secondary Outcome: Number of Participants by Participant's Assessment of Global Aesthetic Improvement Score Categories as Measured by the 5-point GAIS
Description: The participant assessed their global aesthetic improvement using the GAIS 5-point scale where: 2=Much Improved, 1= Improved, 0=No Change, -1=Worse, -2=Much Worse. The number of participants in each score response category at each timepoint is reported.
Time Frame: Day 30, Months 3, 6, and 12
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Juvéderm® VOLIFT™ With Lidocaine
Number analyzed (Participants) | 59
Participants
  Day 30: 2=Much Improved | 32
  Day 30: 1=Improved | 25
  Day 30: 0=No Change | 1
  Day 30: -1=Worse | 1
  Day 30: -2=Much Worse | 0
  Month 3: number analyzed (Participants) | 52
  Month 3: 2=Much Improved | 28
  Month 3: 1=Improved | 21
  Month 3: 0=No Change | 3
  Month 3: -1=Worse | 0
  Month 3: -2=Much Worse | 0
  Month 6: number analyzed (Participants) | 51
  Month 6: 2=Much Improved | 15
  Month 6: 1=Improved | 34
  Month 6: 0=No Change | 2
  Month 6: -1=Worse | 0
  Month 6: -2=Much Worse | 0
  Month 12: number analyzed (Participants) | 36
  Month 12: 2=Much Improved | 6
  Month 12: 1=Improved | 25
  Month 12: 0=No Change | 5
  Month 12: -1=Worse | 0
  Month 12: -2=Much Worse | 0

6. Secondary Outcome: Number of Participants by Assessment of Natural Look of Their Lips Score Category as Measured by a 5-point Likert Scale
Description: The participant assessed the natural look of their lips using a 5-point Likert scale where: 0=Not at All to 4=Very Much. The number of participants in each score response category at each timepoint is reported.
Time Frame: Day 30, Months 3, 6, and 12
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Juvéderm® VOLIFT™ With Lidocaine
Number analyzed (Participants) | 59
Participants
  Day 30: 0=Not at all | 0
  Day 30: 1 | 0
  Day 30: 2=Somewhat | 3
  Day 30: 3 | 18
  Day 30: 4=Very much | 38
  Day 30: Missing | 0
  Month 3: number analyzed (Participants) | 52
  Month 3: 0=Not at all | 0
  Month 3: 1 | 0
  Month 3: 2=Somewhat | 0
  Month 3: 3 | 15
  Month 3: 4=Very much | 37
  Month 3: Missing | 0
  Month 6: number analyzed (Participants) | 51
  Month 6: 0=Not at all | 0
  Month 6: 1 | 0
  Month 6: 2=Somewhat | 1
  Month 6: 3 | 20
  Month 6: 4=Very much | 30
  Month 6: Missing | 0
  Month 12: number analyzed (Participants) | 36
  Month 12: 0=Not at all | 0
  Month 12: 1 | 0
  Month 12: 2=Somewhat | 4
  Month 12: 3 | 5
  Month 12: 4=Very much | 26
  Month 12: Missing | 1

7. Secondary Outcome: Number of Participants by Assessment of Natural Feel of Their Lips Score Category as Measured by a 5-point Likert Scale
Description: The participant assessed the natural feel of their lips using a 5-point Likert scale where: 0=Not at All to 4=Very Much. The number of participants in each score response category at each timepoint is reported.
Time Frame: Day 30, Months 3, 6, and 12
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Juvéderm® VOLIFT™ With Lidocaine
Number analyzed (Participants) | 59
Participants
  Day 30: 0=Not at all | 1
  Day 30: 1 | 0
  Day 30: 2=Somewhat | 5
  Day 30: 3 | 21
  Day 30: 4=Very much | 32
  Month 3: number analyzed (Participants) | 52
  Month 3: 0=Not at all | 0
  Month 3: 1 | 0
  Month 3: 2=Somewhat | 1
  Month 3: 3 | 17
  Month 3: 4=Very much | 34
  Month 6: number analyzed (Participants) | 51
  Month 6: 0=Not at all | 0
  Month 6: 1 | 0
  Month 6: 2=Somewhat | 2
  Month 6: 3 | 21
  Month 6: 4=Very much | 28
  Month 12: number analyzed (Participants) | 36
  Month 12: 0=Not at all | 0
  Month 12: 1 | 0
  Month 12: 2=Somewhat | 4
  Month 12: 3 | 4
  Month 12: 4=Very much | 28

8. Secondary Outcome: Number of Participants by Investigator's Assessment of Product Smoothness Score Categories as Measured by a 5-point Scale
Description: The Investigator evaluated the smoothness of product using a 5-point scale where: 0=Lumpy/Grainy, 1=Faintly Smooth, 2=Somewhat Smooth, 3= Smooth, and 4=Very Smooth. The number of participants in each score response category at each timepoint is reported.
Time Frame: Day 30, Months 3, 6, and 12
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Juvéderm® VOLIFT™ With Lidocaine
Number analyzed (Participants) | 59
Participants
  Day 30: 0=Lumpy/Grainy | 0
  Day 30: 1=Faintly Smooth | 1
  Day 30: 2=Somewhat Smooth | 1
  Day 30: 3=Smooth | 22
  Day 30: 4=Very Smooth | 35
  Month 3: number analyzed (Participants) | 52
  Month 3: 0=Lumpy/Grainy | 0
  Month 3: 1=Faintly Smooth | 0
  Month 3: 2=Somewhat Smooth | 3
  Month 3: 3=Smooth | 14
  Month 3: 4=Very Smooth | 35
  Month 6: number analyzed (Participants) | 51
  Month 6: 0=Lumpy/Grainy | 0
  Month 6: 1=Faintly Smooth | 0
  Month 6: 2=Somewhat Smooth | 1
  Month 6: 3=Smooth | 17
  Month 6: 4=Very Smooth | 33
  Month 12: number analyzed (Participants) | 36
  Month 12: 0=Lumpy/Grainy | 0
  Month 12: 1=Faintly Smooth | 1
  Month 12: 2=Somewhat Smooth | 2
  Month 12: 3=Smooth | 0
  Month 12: 4=Very Smooth | 33

9. Secondary Outcome: Number of Participants by Investigator's Assessment of Dynamic Lip Lines Upon Animation Score Categories
Description: The investigator evaluated the improvement of the participant's dynamic lip lines upon animation using a 4-point scale where: 0=Worse, 1=No Change, 2=Improved, 3=Much Improved. The number of participants in each score response category at each timepoint is reported.
Time Frame: Day 30, Months 3, 6, and 12
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Juvéderm® VOLIFT™ With Lidocaine
Number analyzed (Participants) | 59
Participants
  Day 30: 0=Worse | 0
  Day 30: 1=No Change | 2
  Day 30: 2=Improved | 30
  Day 30: 3=Much Improved | 27
  Month 3: number analyzed (Participants) | 52
  Month 3: 0=Worse | 0
  Month 3: 1=No Change | 2
  Month 3: 2=Improved | 28
  Month 3: 3=Much Improved | 22
  Month 6: number analyzed (Participants) | 51
  Month 6: 0=Worse | 0
  Month 6: 1=No Change | 6
  Month 6: 2=Improved | 26
  Month 6: 3=Much Improved | 19
  Month 12: number analyzed (Participants) | 36
  Month 12: 0=Worse | 0
  Month 12: 1=No Change | 10
  Month 12: 2=Improved | 20
  Month 12: 3=Much Improved | 6

ADVERSE EVENTS:
Time Frame: First dose of study treatment to the end of the study (Up to Month 12)
Description: Safety Analysis Set included all participants who were consented and enrolled into this study and were treated with the investigational product Juvéderm® VOLIFT™ with Lidocaine.
Arm/Group | Juvéderm® VOLIFT™ With Lidocaine
All-Cause Mortality (participants affected / at risk) | 0/60
Serious Adverse Events (participants affected / at risk) | 0/60
Other Adverse Events (participants affected / at risk) | 0/60

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2019-10-10): https://cdn.clinicaltrials.gov/large-docs/28/NCT03796728/Prot_000.pdf
  • Statistical Analysis Plan (2019-10-10): https://cdn.clinicaltrials.gov/large-docs/28/NCT03796728/SAP_001.pdf